CLINICAL TRIAL: NCT06213922
Title: Prevalence of and Risk Factors of Obesity in School Children and Adolescents in Nag Hammadi City.
Brief Title: Prevalence of and Risk Factors of Obesity in School Children and Adolescents in Nag Hammadi City. 300 Participants.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Doaa Hagoug Ahmed, Nag Hammadi health administration, Sohag University
Other Study IDs: Soh-Med-23-11-05MS
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Obesity, Adolescent
Keywords: Body mass index
MeSH Terms: conditions — Pediatric Obesity | interventions — Eating

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescent
  Interventions: Behavioral: Food intake

INTERVENTIONS:
Behavioral: Food intake — Fast food

SUMMARY:
Searching for obese children who's body mass index is above normal range and risk factors in children and adolescents in Nag Hammadi city

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents 12to18years.

Exclusion Criteria:

* children younger than12 years and who have special conditions as deaf.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Community study
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in dietary habits | 6 months

IPD SHARING:
Plan to Share IPD: No